CLINICAL TRIAL: NCT07237048
Title: Effect of Oral Minocycline in Patients With Acute Stroke - a Randomized, Open Label, Prospective Trial
Brief Title: Minocycline in Stroke Study at Maimonides
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joyce Chen (Other)
Responsible Party: Sponsor-Investigator, Joyce Chen, Clinical Data Analyst, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-05-01-MMC; Internal Stroke Research Funds (Other Grant/Funding Number: Internal Stroke Research Funds)
Record Dates: First submitted 2025-10-23; First posted 2025-11-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Ischemia Stroke; Hemorrhagic Strokes; Mortality; Morbidity; Cerebrovascular Accident (Stroke); Intracerebral Haemorrhage (ICH)
Keywords: Minocycline; Acute Stroke; Neuroprotection; Ischemic Stroke; Hemorrhagic Stroke; NIH Stroke Scale; Modified Rankin Scale (mRS); Stroke Recovery; Stroke Treatment; Stroke Outcomes; Morbidity; Mortality; Intravenous Thrombolysis; Mechanical Thrombectomy; Hemorrhagic Transformation; Oral antibiotic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebral Hemorrhage; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Randomized, open label, prospective
Who Masked: Outcomes Assessor
Masking Description: This is an outcome assessor-blinded study. Independent outcome assessor will contact participants and obtain primary outcome measures of mRS *(Modified Rankin Scale) * and NIHSS *(National Institute of Stroke Scale) * without the knowledge of participants group assignment/treatment received to reduce the bias and improve validity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Stroke Care without Minocycline (No Intervention): 582 Patients in this arm will receive standard stroke care, No Minocycline will be given
- Standard Stroke Care with Minocycline (Experimental): 582 patients in the Minocycline arm will receive Minocycline 200 mg every 24 hours for five days with standard stroke care
  Interventions: Drug: Minocycline 200mg

INTERVENTIONS:
Drug: Minocycline 200mg — Minocycline 200 mg every 24 hours for five days to be initiated within 24hr of stroke onset.
  Other Names: Minocin; Minocycline hydrochloride
  Arms: Standard Stroke Care with Minocycline

SUMMARY:
The goal of this study is to determine if Minocycline, when added to standard care, can improve survival and functional outcomes in patients with moderate acute stroke (ischemic or hemorrhagic) aged 18 years and older.

The main questions it aims to answer are:

1. Does Minocycline improve *National Institutes of Health Stroke Scale* (NIHSS) scores at hospital discharge and 90 days post-stroke?
2. Does Minocycline reduce stroke-related disability, all-cause in hospital mortality (mRS -*Modified Rankin Scale* = 6) and at 90 days besides reducing brain bleeding complications compared to standard care?

Researchers will compare patients receiving oral Minocycline plus standard care to those receiving standard care only to see if Minocycline leads to better neurological outcomes and lower mortality.

Participants will:

1. Be randomly assigned by block to receive either:

   Minocycline 200 mg orally once daily for five days within 24 hours from symptoms onset + Standard Care, or Standard Care only
2. Undergo neurological assessments using NIHSS *National Institutes of Health Stroke Scale* and Modified Rankin Scale (mRS) at admission, discharge, 30 days post-stroke, 90 days post-stroke
3. Be monitored for: a) hemorrhagic transformation of ischemic strokes; b) Adverse events and mortality outcomes; c) Safety and efficacy signals through interim analyses

NIHSS: *National Institutes of Health Stroke Scale*, which is stroke severity scale,

mRS: *Modified Rankin Scale*, which is stroke disability scale

DETAILED DESCRIPTION:
Stroke is a major cause of death and disability in the United States. While treatments such as clot-busting drugs (tPA or TNK) and thrombectomy can help some patients with ischemic strokes, there are limited options for protecting the brain after a stroke. Minocycline is a low-cost antibiotic that may have protective effects on the brain due to its anti-inflammatory and neuroprotective properties.

At Maimonides Medical Center, we have used Minocycline for all eligible patients with acute strokes in clinical practice until March 2019, Studies found that Minocycline was associated with better stroke outcomes and lower death rates, especially in patients with moderate stroke severity. However, no large, randomized trial has yet confirmed its benefits.

This study will prospectively enroll 1,164 adults with moderate stroke (National Institutes of Health Stroke Scale 5-20) within 24 hours of symptom onset. Participants will be assigned by block randomization to receive either:

Minocycline 200 mg orally once daily for 5 days + standard stroke care, or Standard stroke care alone.

The study will measure stroke severity (using the *NIHSS*- National Institutes of Health Stroke Scale) and disability (using the mRS - *modified Rankin Scale*) at hospital discharge, 30 days, and 90 days. It will also monitor for death and any bleeding complications in the brain.

The goal is to see whether Minocycline, in addition to usual care, can safely improve recovery and survival in people with acute stroke. The results could help guide future stroke treatment nationwide.

NIHSS: *National Institutes of Health Stroke Scale*, is stroke severity scale, mRS: *Modified Rankin Scale*, is stroke disability scale, WHO: *World Health Organization*

ELIGIBILITY:
* Inclusion criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age >/=18
2. NIHSS 5-20 *National Institutes of Health Stroke Scale*
3. Acute onset neurological deficit consistent with acute ischemic stroke or on imaging consistent with acute ischemia as defined by WHO *(World Health Organization) * guidelines or acute onset of neurological deficits with intracerebral Hemorrhage on imaging consistent with intracerebral bleed
4. The onset of neurological symptoms less than 24 hours

   * Exclusion criteria

An individual who meets any of the following criteria is excluded from participation in this study:

1. Clinically stroke is not suspected
2. Allergic to the Tetracycline group of medications or Intolerance to Minocycline
3. Pregnancy or suspected pregnancy or breastfeeding
4. Previous history of intolerance to Minocycline
5. Acute or chronic renal failure (stage III with GFR *(Glomerular Filtration Rate) * or Creatinine threshold)
6. Any patients with contraindications to undergo CT (Computed Tomography) / MRI (Magnetic Resonance Imaging)
7. Life expectancy less than one year or severe co-morbidities or comfort measure only (CMO) on admission
8. Pre-existing infectious disease requiring antibiotics
9. Inability to tolerate enteral medications/feeds
10. Patient/ family refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in National Institutes of Health Stroke Scale (NIHSS) Score at Day 7 post stroke | At day 7 after stroke onset
  The NIHSS score will be assessed at Day 7 post-stroke to measure neurological impairment and recovery. The primary outcome is the difference in NIHSS scores between the Minocycline plus standard care group and the standard care alone group.
Change in National Institutes of Health Stroke Scale (NIHSS) Score at 90 days (+/- 7 days) post-stroke | At 90 days (+/- 7 days) after stroke onset
  The NIHSS score will be assessed 90 days (+/- 7 days) post-stroke to measure neurological impairment and recovery. The primary outcome is the difference in NIHSS scores between the Minocycline plus standard care group and the standard care alone group.

SECONDARY OUTCOMES:
NIHSS Score at 30 Days Post-Stroke | up to 30 days after stroke onset
  NIHSS scores will be assessed at 30 days (+/- 7 days) post-stroke to evaluate intermediate neurological recovery in both treatment arms.
Rate of Hemorrhagic Transformation of Ischemic Strokes | 22-36 hours post treatment
  The incidence of hemorrhagic transformation in ischemic stroke patients treated with IV thrombolytics and/or thrombectomy will be assessed during hospitalization using ECASS ( European Cooperative Acute Stroke Study) II/III criteria via follow-up CT or MRI imaging.
All-Cause Mortality (mRS = 6) | Up to 90 days (±7 days) after stroke onset
  Mortality rates will be measured at Day 7, 30 days (+/- 7 days), and 90 days (+/- 7 days) post-stroke in both treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Qingliang T. Wang, MD, PhD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT07237048/Prot_SAP_000.pdf